CLINICAL TRIAL: NCT07080138
Title: Research on the Psychological Status of Patients With HIV-1 Infection
Status: Not yet recruiting | Type: Observational
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: YXLL-2024-162
Record Dates: First submitted 2025-07-14; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2024-09

CONDITIONS: HIV-1-infection; Anxiety Depression
MeSH Terms: interventions — bictegravir; dolutegravir; abacavir, dolutegravir, and lamivudine drug combination; albuvirtide; Lamivudine; elvitegravir; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Emtricitabine; lamivudine, zidovudine drug combination; Raltegravir Potassium; Rilpivirine; abacavir; efavirenz; Lopinavir; Nevirapine; Tenofovir; Zidovudine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Gender, Age, therapeutic regimen, medication time, Clinical patient blood, PsychoSocial Index, PSQI, and MemTrax.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group INSTI: Treated by INSTI
  Interventions: Drug: All kinds of INSTI medications
- Group CONV: Treated by Conventional medicines
  Interventions: Drug: All kinds of conventional medications

INTERVENTIONS:
Drug: All kinds of INSTI medications — All kinds of INSTI medications, such as Bictegravir/Emtricitabine/Tenofovir alafenamide Fumarate, Dolutegravir/Emtricitabine/Tenofovir alafenamide Fumarate for PLWH
  Other Names: Bictegravir/Emtricitabine/Tenofovir alafenamide Fumarate; Dolutegravir/Emtricitabine/Tenofovir alafenamide Fumarate; Abacavir/Dolutegravir/Lamivudine; Albuvirtide; Dolutegravir; Dolutegravir/Lamivudine; Elvitegravir/Cobicistat/Emtricitabine/Tenofovir alafenamide Fumarate; Emtricitabine/Tenofovir; Emtricitabine/Tenofovir alafenamide Fumarate; Enovirin; Lamivudine/Zidovudine; Raltegravir; Rilpivirine
  Groups: Group INSTI
Drug: All kinds of conventional medications — All kinds of conventional medications, such as Abacavir, Efavirenz for PLWH
  Other Names: Abacavir; Efavirenz; Emtricitabine; Lamivudine; Lopinavir/Ritonavir; Nevirapine; Tenofovir; Tenofovir alafenamide Fumarate; Zidovudine
  Groups: Group CONV

SUMMARY:
The goal of this observational study is to investigate the neuropsychological states of People Living With HIV(PLWH), the prevalence of social and psychological stress adaptation overload and poor episodic memory in PLWH. The main questions it aims to observe are: to observe the prevalence of psychopathic states in PLWH with different viral loads and to compare the effects of different treatments on the prevalence of psychopathic states in PLWH. It is helpful to understand the mental health burden faced by PLWH in China, to improve clinicians' awareness of PLWH's mental and psychological state, and formulate targeted psychological support, treatment and nursing programs.

DETAILED DESCRIPTION:
Our research is a prospective cohort of PLWH, mainly observing the differences in the prevalence of AO among different treatment strategies; Secondly, observe: ① The changes of neuropsychological symptoms such as newly diagnosed PLWH, AO, and Poor EM compared with the baseline; ② Changes in neuropsychological symptoms such as PLWH, AO, and Poor EM after treatment with different treatment regimens compared to the baseline; ③ For PLWH at different stages, after half a year of treatment, the changes of neuropsychological symptoms such as PLWH, AO, and Poor EM compared with the baseline; ④ Changes in Interpersonal Stress, Work Stress and Daily Stress conditions of PLWH compared with the baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis: PLWH can be diagnosed if one of the following three items is met according to the Chinese AIDS Diagnosis and Treatment Guidelines (2021):

   ① HIV antibody screening test positive and HIV supplementation test positive (antibody supplementation test positive or nucleic acid qualitative test positive or nucleic acid quantification>5000 copies/mL);

   ② Has a history of epidemiology or clinical manifestations related to AIDS, tested positive for HIV nucleic acid twice;

   ③ HIV isolation test positive;
2. Receive treatment at the hospital participating in the study; Age range: 18-80 years old, male or female not limited;
3. Patients who are willing to participate in this clinical study and sign the informed consent form for this study.

Exclusion Criteria:

Individuals who meet any of the following criteria are not eligible to participate in this study:

1. Pregnant or lactating women; Men and women who are preparing for natural conception or artificial assisted reproduction;
2. Severe aphasia, physical disability, or any other non neuropsychological factors that may hinder the completion of the assessment;
3. is currently involved in other research;
4. Having a tendency towards violence may endanger the safety of others.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People Living With HIV
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The prevalence of AO among different treatment strategies | 2025.8-2026.7
  Observe the differences in the prevalence of AO in PLWH under different treatment strategies

SECONDARY OUTCOMES:
The changes of Poor EM after the treatment of newly diagnosed PLWH | 2025.8-2026.7
  The changes of Poor EM neuropsychological symptoms in newly diagnosed PLWH compared with the baseline under different treatment regimens

OTHER OUTCOMES:
The changes of Poor EM after the treatment of treated PLWH | 2025.8-2026.7
  The changes of Poor EM neuropsychological symptoms in treated diagnosed PLWH compared with the baseline under different treatment regimens
The changes in Interpersonal Stress, Work Stress and Daily Stress conditions of PLWH | 2025.8-2026.7
  The changes in Interpersonal Stress, Work Stress and Daily Stress conditions of PLWH compared with the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Xingyu Li, doctor, Principal Investigator — Shanxi Bethune Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Niu L, Luo D, Liu Y, Silenzio VM, Xiao S. The Mental Health of People Living with HIV in China, 1998-2014: A Systematic Review. PLoS One. 2016 Apr 15;11(4):e0153489. doi: 10.1371/journal.pone.0153489. eCollection 2016. PMID 27082749
- [Background] Bing EG, Burnam MA, Longshore D, Fleishman JA, Sherbourne CD, London AS, Turner BJ, Eggan F, Beckman R, Vitiello B, Morton SC, Orlando M, Bozzette SA, Ortiz-Barron L, Shapiro M. Psychiatric disorders and drug use among human immunodeficiency virus-infected adults in the United States. Arch Gen Psychiatry. 2001 Aug;58(8):721-8. doi: 10.1001/archpsyc.58.8.721. PMID 11483137
- [Background] Elendu C, Aguocha CM, Okeke CV, Okoro CB, Peterson JC. HIV-related neurocognitive disorders: Diagnosis, Treatment, and Mental Health Implications: A Review. Medicine (Baltimore). 2023 Oct 27;102(43):e35652. doi: 10.1097/MD.0000000000035652. PMID 37904369
- [Background] Remien RH, Stirratt MJ, Nguyen N, Robbins RN, Pala AN, Mellins CA. Mental health and HIV/AIDS: the need for an integrated response. AIDS. 2019 Jul 15;33(9):1411-1420. doi: 10.1097/QAD.0000000000002227. PMID 30950883
- [Background] Guidi J, Lucente M, Sonino N, Fava GA. Allostatic Load and Its Impact on Health: A Systematic Review. Psychother Psychosom. 2021;90(1):11-27. doi: 10.1159/000510696. Epub 2020 Aug 14. PMID 32799204
- [Background] Bobba-Alves N, Juster RP, Picard M. The energetic cost of allostasis and allostatic load. Psychoneuroendocrinology. 2022 Dec;146:105951. doi: 10.1016/j.psyneuen.2022.105951. Epub 2022 Oct 8. PMID 36302295
- [Background] Palego L, Giannaccini G, Betti L. Neuroendocrine Response to Psychosocial Stressors, Inflammation Mediators and Brain-periphery Pathways of Adaptation. Cent Nerv Syst Agents Med Chem. 2021;21(1):2-19. doi: 10.2174/1871524920999201214231243. PMID 33319677
- [Background] Sonino N, Fava GA, Lucente M, Guidi J. Allostatic Load and Endocrine Disorders. Psychother Psychosom. 2023;92(3):162-169. doi: 10.1159/000530691. Epub 2023 May 30. PMID 37253338
- [Background] Eory A, Bekesi D, Eory A, Rozsa S. Physical Exercise as a Resilience Factor to Mitigate COVID-Related Allostatic Overload. Psychother Psychosom. 2021;90(3):200-206. doi: 10.1159/000514331. Epub 2021 Mar 10. PMID 33691321
- [Background] Zhao S, Shibata K, Hellyer PJ, Trender W, Manohar S, Hampshire A, Husain M. Rapid vigilance and episodic memory decrements in COVID-19 survivors. Brain Commun. 2022 Jan 19;4(1):fcab295. doi: 10.1093/braincomms/fcab295. eCollection 2022. PMID 35128398
- [Background] Ripamonti E, Clerici M. The association of memory disorders and chronic HIV disease in the antiretroviral therapy era: a systematic literature review. HIV Med. 2020 Jan;21(1):9-20. doi: 10.1111/hiv.12793. Epub 2019 Oct 11. PMID 31603624
- [Background] Ji J, Zhang Y, Ma Y, Jia L, Cai M, Li Z, Zhang T, Guo C. People who living with HIV/AIDS also have a high prevalence of anxiety disorders: a systematic review and meta-analysis. Front Psychiatry. 2024 Feb 6;15:1259290. doi: 10.3389/fpsyt.2024.1259290. eCollection 2024. PMID 38380124
- [Background] Bhatia MS, Munjal S. Prevalence of Depression in People Living with HIV/AIDS Undergoing ART and Factors Associated with it. J Clin Diagn Res. 2014 Oct;8(10):WC01-4. doi: 10.7860/JCDR/2014/7725.4927. Epub 2014 Oct 20. PMID 25478433
- [Background] Regan M, Muhihi A, Nagu T, Aboud S, Ulenga N, Kaaya S, Fawzi MCS, Yousafzai AK, Mugusi F, Fawzi WW, Saxena S, Koenen K, Sudfeld CR. Depression and Viral Suppression Among Adults Living with HIV in Tanzania. AIDS Behav. 2021 Oct;25(10):3097-3105. doi: 10.1007/s10461-021-03187-y. Epub 2021 Feb 17. PMID 33598866
- [Background] Ruhanya V, Jacobs GB, Naidoo S, Paul RH, Joska JA, Seedat S, Nyandoro G, Engelbrecht S, Glashoff RH. Impact of Plasma IP-10/CXCL10 and RANTES/CCL5 Levels on Neurocognitive Function in HIV Treatment-Naive Patients. AIDS Res Hum Retroviruses. 2021 Sep;37(9):657-665. doi: 10.1089/AID.2020.0203. Epub 2021 Feb 17. PMID 33472520
- [Background] Levy ME, Monroe AK, Horberg MA, Benator DA, Molock S, Doshi RK, Powers Happ L, Castel AD. Pharmacologic Treatment of Psychiatric Disorders and Time With Unsuppressed HIV Viral Load in a Clinical HIV Cohort. J Acquir Immune Defic Syndr. 2019 Nov 1;82(3):329-341. doi: 10.1097/QAI.0000000000002138. PMID 31356466
- [Result] Stadtler H, Shaw G, Neigh GN. Mini-review: Elucidating the psychological, physical, and sex-based interactions between HIV infection and stress. Neurosci Lett. 2021 Mar 16;747:135698. doi: 10.1016/j.neulet.2021.135698. Epub 2021 Feb 1. PMID 33540057